CLINICAL TRIAL: NCT02361151
Title: Enhancing Parent-Child Communication and Promoting Physical Activity and Healthy Eating Through Mobile Technology: the mFIT Study (Motivating Families With Interactive Technology)
Brief Title: The mFIT Study (Motivating Families With Interactive Technology)
Acronym: mFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Advisor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00038855
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TECH (standard program) (Active Comparator): Receive 3-month healthy eating and physical activity intervention delivered via email newsletters and mobile apps plus self-monitoring with paper records; based on standard behavior change recommendations and materials (e.g., Diabetes Prevention Program)
  Intervention: remotely-delivered evidence-based intervention to support healthy eating and physical activity; use of supporting app-based games and activities and self-monitoring.
  Interventions: Behavioral: TECH
- TECH+ (enhanced program) (Experimental): Receive 3-month family-based healthy eating and physical activity intervention delivered via email newsletters and mobile apps plus self-monitoring with special study website
  Intervention: remotely-delivered evidence-based intervention to support healthy eating and physical activity; use of supporting app-based games and activities; enhanced self-monitoring and family activities via special study website
  Interventions: Behavioral: TECH+

INTERVENTIONS:
Behavioral: TECH — Weekly newsletter with health information, mobile apps, and self-monitoring materials
  Arms: TECH (standard program)
Behavioral: TECH+ — Weekly newsletter with health information, mobile apps, and self-monitoring materials along with theory-based mobile web intervention
  Arms: TECH+ (enhanced program)

SUMMARY:
The high rates of childhood obesity in the US demand innovative and cost-effective weight gain prevention tools; mobile applications (apps) represent one such solution. Using a randomized design, the mFIT study tests the effectiveness of using commercially available apps and a physical activity (PA) monitoring device (Tech, n=50 parent-child dyads) compared to the apps and PA device plus a mobile website and theory-based family intervention that encourages increased parent-child communication about PA and healthy eating as well as family behavior change (Tech+, n=50 parent-child dyads).

DETAILED DESCRIPTION:
Objectives and Significance. Finding scalable and engaging ways to disseminate obesity treatment and prevention for children has been challenging. Mobile applications (apps) are an engaging way to involve children in health behavior changes, capitalizing on the portability and affordability of delivering health information via mobile devices and the opportunity to use gaming to make health information entertaining. Previous research by our team, including a systematic review of commercially available mobile apps for family weight loss, physical activity, and healthy eating as well as a pilot test of commercially available apps and physical activity monitoring devices with parent-child dyads, revealed significant gaps in the available mobile tools. The proposed study will test the effectiveness of using commercially available apps and a physical activity monitoring device (Tech) compared to the apps and physical activity device plus a mobile website and theory-based family intervention that encourages increased parent-child communication about physical activity and healthy eating and family behavior change (Tech+). The two programs will be administered remotely via email, mobile apps, and a mobile website to parent-child dyads (child 9-12 years old), using over a 3-month intervention period. Parent-child dyads will be randomized to the two behavioral interventions: Tech (50 dyads) or Tech+ (50 dyads). Our proposed research has two aims:

Aim 1: Test the effectiveness of an evidence-based mobile intervention with enhanced parent/child communication (Tech+) versus commercially available products (physical activity and healthy eating apps, physical activity device) alone (Tech) for improvements in physical activity and healthy eating in parents and children.

Aim 2: Examine the impacts of evidence-based family intervention on parent-child relationship quality and communication about physical activity and healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* Participants must include 1 child (age 9-12) and their parent or guardian
* Parent not currently meeting physical activity guidelines (participants will be eligible if they currently engage in aerobic activities for less than 2 hours and 30 minutes/week and strength training <2 days/week)
* Own and use a smartphone and/or a tablet with a data plan (e.g., iPhone, iPad)
* Live in the same household as the child
* Are willing to be randomized to one of the two intervention groups
* Willing and able to be physically active

Exclusion Criteria:

* Has a psychiatric disease, drug or alcohol dependency, or uncontrolled thyroid condition
* Has an eating disorder
* Currently participating in a weight loss program or taking weight loss medications
* Has a major chronic diseases, including: heart disease, past incidence of stroke, uncontrolled diabetes

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Bouts of moderate-to-vigorous physical activity (via accelorometers) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Turner-McGrievy, PhD, MS, RD, Study Chair — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States